CLINICAL TRIAL: NCT01143337
Title: A Multicenter Randomized, Double-blind, Placebo-controlled Study of MP-435 in Combination With MTX in Patients With Rheumatoid Arthritis - Exploratory Study
Brief Title: Efficacy and Safety Study of MP-435 in Combination With Methotrexate (MTX) in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-435-J04
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dose1
  Interventions: Drug: MP-435(dose1) + Methotrexate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo + Methotrexate

INTERVENTIONS:
Drug: MP-435(dose1) + Methotrexate — MP-435 dose1 + stable weekly dose of Methotrexate
  Arms: 1
Drug: Placebo + Methotrexate — Placebo + stable weekly dose of Methotrexate
  Arms: 2

SUMMARY:
The purpose of this study is to determine the Efficacy, Safety, and Pharmacokinetics of MP-435 administered for 12 weeks in subjects with rheumatoid arthritis (RA) on stable doses of Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RA according to the diagnostic criteria of the American College of Rheumatology (ACR) (revised in 1987) for at least 6 months.
* Subjects who inadequately response for stable dose of MTX.

Exclusion Criteria:

* Patients with Class IV functional activity by the Steinbrocker's scale.
* Patients who have received a biological agent in the past.
* Patients who have other rheumatic diseases, or who have other diseases with joint symptoms.
* Patients with severe or uncontrolled endocrine, psychiatric, cardiac, hematological, pulmonary, hepatic, kidney, gastrointestinal, or thyroid disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: MP-435 placebo-matching tablets, orally, twice daily. And stable dose (6-8 mg/week) Methotrexate(MTX) were administered as background therapy.
- MP-435 100mg BID: MP-435 100mg, orally, twice daily. And stable dose (6-8 mg/week) MTX were administered as background therapy.
- MP-435 400mg BID: MP-435 400mg, orally, twice daily. And stable dose (6-8 mg/week) MTX were administered as background therapy.
Period: Overall Study
Arm/Group | Placebo | MP-435 100mg BID | MP-435 400mg BID
Started | 49 | 50 | 13
Completed | 39 | 39 | 1 (Frequency of this arm AE was higher than assumption before study initiation.)
Not Completed | 10 | 11 | 12
Not completed — Adverse Event | 3 | 9 | 5
Not completed — Lack of Efficacy | 6 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other reason | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- MP-435 100mg BID: MP-435 100mg, orally, twice daily. And stable dose (6-8 mg/week) MTX were administered as background therapy.
  MP-435 400mg:
  There were 13 patients who randomized 400 mg bid group when they were discontinued dosing. At this point, it was found that there were Four patients who increased ALT more than three times of upper limit of normal in this dosing group. Therefore, patients who randomized to this dosing group were discontinued and also new inclusion was stopped in this point.
  Primary analysis of this study result was Par Protocol Set ( PPS ). Because examination for 400 mg bid group was discontinued, this arm data was excluded from PPS analysis.
- Total: Total of all reporting groups
Arm/Group | Placebo | MP-435 100mg BID | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Customized [Number; unit: participants]
  < 40 years | 5 | 8 | 13
  40 - 50 years | 9 | 7 | 16
  50 - 60 years | 13 | 13 | 26
  60 - 70 years | 15 | 12 | 27
  ≧ 70 years | 4 | 7 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 (ACR 20) Response
Description: ACR 20 response is a decrease of at least 20 per cent in both tender and swollen joint count [TJC and SJC] and in 3 to 5 assessments (participant's assessment of pain visual analog scale [VAS] with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; Health Assessment Questionnaire [HAQ-DI]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; C-reactive protein[CRP]).
Time Frame: Week 2, 4, 6, 8, 12, LOCF (Week 12 or discontinuation time)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MP-435 100mg BID
Number analyzed (Participants) | 46 | 47
percentage of participants
  Week 2 | 10.9 [3.6 to 23.6] | 19.1 [9.1 to 33.3]
  Week 4 | 24.4 [12.9 to 39.5] | 39.1 [25.1 to 54.6]
  Week 6 | 23.3 [11.8 to 38.6] | 39.0 [24.2 to 55.5]
  Week 8 | 34.9 [21.0 to 50.9] | 45.0 [29.3 to 61.5]
  Week 12 | 39.5 [24.0 to 56.6] | 39.5 [24.0 to 56.6]
  LOCF (Week 12 or discontinuation time) | 34.8 [21.4 to 50.2] | 42.6 [28.3 to 57.8]

2. Secondary Outcome: Percentage of Participants Achieving ACR 50 Response
Description: ACR 50 response is a decrease of at least 50 per cent in both tender and swollen joint count and in 3 to 5 assessments (participant's assessment of pain VAS with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; HAQ-DI: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; CRP).
Time Frame: Week 2, 4, 6, 8, 12, LOCF (Week 12 or discontinuation time)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MP-435 100mg BID
Number analyzed (Participants) | 46 | 47
percentage of participants
  Week 2 | 4.3 [0.5 to 14.8] | 2.1 [0.1 to 11.3]
  Week 4 | 8.9 [2.5 to 21.2] | 4.3 [0.5 to 14.8]
  Week 6 | 7.0 [1.5 to 19.1] | 12.2 [4.1 to 26.2]
  Week 8 | 9.3 [2.6 to 22.1] | 17.5 [7.3 to 32.8]
  Week 12 | 13.2 [4.4 to 28.1] | 15.8 [6.0 to 31.1]
  LOCF (Week 12 or discontinuation time) | 13.0 [4.9 to 26.3] | 14.9 [6.2 to 28.3]

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 (ACR 70) Response
Description: ACR 70 response is a decrease of at least 70 per cent in both tender and swollen joint count and in 3 to 5 assessments (participant's assessment of pain VAS with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; HAQ-DI: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; CRP).
Time Frame: Week 2, 4, 6, 8, 12, LOCF (Week 12 or discontinuation time)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MP-435 100mg BID
Number analyzed (Participants) | 46 | 47
percentage of participants
  Week 2 | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.5]
  Week 4 | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 7.7]
  Week 6 | 2.3 [0.1 to 12.3] | 0.0 [0.0 to 8.6]
  Week 8 | 2.3 [0.1 to 12.3] | 0.0 [0.0 to 8.8]
  Week 12 | 2.6 [0.1 to 13.8] | 2.6 [0.1 to 13.8]
  LOCF (Week 12 or discontinuation time) | 2.2 [0.1 to 11.5] | 4.3 [0.5 to 14.5]

4. Secondary Outcome: Changes From the Pretreatment Values in the Disease Activity Score (DAS) 28, and ACR Components
Description: DAS28 (CRP) is calculated using TJC, SJC C-Reactive Protein ( CRP in mg/dL ), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.36 x log (CRP+1) + 0.014 x Global Assessment of Arthritis + 0.96 where 28 joints are examined and a lower score indicates less disease activity.
  DAS28 (ESR) is calculated using TJC, SJC erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x log (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
  A negative change score indicates improvement. Higher score indicated more disease activity. DAS28 =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate disease activity, >5.1 implied high disease activity.
Time Frame: LOCF (Week 12 or discontinuation time)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MP-435 100mg BID
Number analyzed (Participants) | 46 | 47
units on a scale
  DAS 28 (CRP) Week 0 | 4.18 (0.80) | 4.41 (0.77)
  DAS 28 (CRP) Week 12 or discontinuation time | 3.48 (1.26) | 3.54 (1.15)
  DAS 28 (ESR) Week 0 | 5.59 (0.82) | 5.8 (0.76)
  DAS 28 (ESR) Week 12 or discontinuation time | 4.87 (1.30) | 4.94 (1.15)

5. Secondary Outcome: Percent Changes From the Pretreatment Values in the Disease Activity Score (DAS) 28, and ACR Components
Description: ACR components are tender joints count (TJC), swollen joints count (SJC), participant assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ-DI]); and C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR).
Time Frame: LOCF (Week 12 or discontinuation time)
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Placebo | MP-435 100mg BID
Number analyzed (Participants) | 46 | 47
percentage of change from baseline
  TJC | 33.72 (52.21) | 36.94 (50.57)
  SJC | 35.74 (91.22) | 44.44 (33.00)
  participant assessment | -2.14 (76.99) | -6.67 (187.29)
  participant global assessment of disease activity | -11.57 (98.92) | 4.53 (128.92)
  physician global assessment of disease activity | 21.6 (43.85) | 33.06 (35.39)
  HAQ-DI | 5.84 (61.48) | 14.78 (49.80)
  CRP | -34.13 (147.17) | -46.01 (150.97)
  ESR | 1.00 (27.76) | -12.01 (46.95)

ADVERSE EVENTS:
Arm/Group | Placebo | MP-435 100mg BID
Serious Adverse Events (participants affected / at risk) | 3/49 | 0/50
Other Adverse Events (participants affected / at risk) | 11/49 | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | MP-435 100mg BID (N=50)
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | MP-435 100mg BID (N=50)
Nasopharyngitis (Infections and infestations) | 7 | 6
Headache (Nervous system disorders) | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 6
Liver function test abnormal (Investigations) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other